CLINICAL TRIAL: NCT03364387
Title: The Clinical Profile, Management and Long-Term Outcomes of Patients With Acute Coronary Syndrome and Myocardial Infarction With Non-obstructive Coronary Arteries in Turkish Population
Brief Title: Myocardial Infarction With Non-obstructive Coronary Arteries in Turkish Population
Acronym: MINOCA-TR
Status: Completed | Type: Observational
Sponsor: Cardiovascular Academy Society, Turkey (Other)
Responsible Party: Sponsor
Other Study IDs: MINOCA-TR
Record Dates: First submitted 2017-11-30; First posted 2017-12-06 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Acute Coronary Syndrome; Myocardial Infarction; Atrial Fibrillation; Diabetes Mellitus
Keywords: Acute Coronary Syndrome; MINOCA; Myocardial Infarction; Atrial Fibrillation
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Atrial Fibrillation; Diabetes Mellitus; MINOCA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fasting venous blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to analyze the Demographics, Clinical Profiles, Management, in-Hospital and Long-Term Outcomes of Patients with Acute Coronary Syndrome Syndrome And Myocardial Infarction with Non-obstructive Coronary Artery Disease.

DETAILED DESCRIPTION:
Acute coronary syndrome is leading causes of death worldwide. Although, >90% of these patients had of culprit coronary lesion, a significant proportion of them had no any angiographic evidence of obstructive coronary arteries. Exact mechanism of the myocardial infarction remains unclear of these patients. However, MI registries have reported that the 5% to %10 of MI patients have no evidence of obstructive coronary artery disease.

There is lack of any data regarding prevalence, demographics, patients' profile, management, and outcome of this clinical entity in Turkish population. This registry aims to obtain these data in Myocardial Infarction with Non-obstructive Coronary Artery Disease patients in Turkish population.

Although there are huge data in this issue from different country and geographic areas, to date no any national data about prevalence, demographics, management and in-hospital outcomes of AF patients who admitting with cute coronary syndrome. With this rationale the registry also aims to obtain demographics, clinical profile, management, and in-hospital outcome of AF in Turkish Acute coronary syndrome population.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 years
2. Evidence of an MI as defined any one of the following criteria:

   Detection of a rise and/or fall of cardiac biomarker values [preferably cardiac troponin (cTn)] with at least one value above the 99th percentile upper reference limit (URL) and with at least one of the following:

   i. Symptoms of ischaemia. ii. New or presumed new signiﬁcant ST-segment-T wave (ST-T) changes or new left bundle branch block (LBBB).

   iii. Development of pathological Q waves in the ECG. iv. Imaging evidence of new loss of viable myocardium or new regional wall motion abnormality.

   v. Identiﬁcation of an intracoronary thrombus by angiography.
3. Invasive diagnostic coronary angiography (IDCA) findings to allow determination of the presence /absence of obstructive coronary artery disease
4. Signed informed consent form to trial participation

Exclusion Criteria:

1. Inability/Refused to provide informed consent
2. Age below 18 years
3. Patients with unstable angina pectoris (ACS without increase and/or decrease of a cardiac biomarker, preferably high-sensitivity cardiac troponin, with at least one value above the 99th percentile of the upper reference limit)
4. Patients refused invasive diagnostic coronary angiography
5. Myocardial infarction associated with revascularization procedures

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study population will consisted patients with acute coronary syndrome undergoing invasive diagnostic coronary angiography.
  Patients will eligible to take part in the study if they will fulfilled the criteria for acute myocardial infarction.
Sampling Method: Probability Sample
Enrollment: 16026 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Composites of Myocardial Infarction, Hospitalization, Revascularization, Death | 12 months
  Re-infarction, Any cause or Cardiovascular Hospitalization or Death

SECONDARY OUTCOMES:
Atrial Fibrillation | 12 months
  Any type of atrial fibrillation
Heart failure | 12 months
  Acute decompensated heart failure with or without cardiogenic shock

CONTACTS AND LOCATIONS:
Locations (1):
- Emin Alioğlu, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No